CLINICAL TRIAL: NCT01995474
Title: Eliminating the Residual Negative Pressure in the EUS-FNA Needle Before Withdrawal Enhances the FNA Cytology Yield
Brief Title: Simple Technique to Improve Diagnostic Yield in EUS-FNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: PRO-00012314
Record Dates: First submitted 2013-04-30; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Lesion Sampled for Cytology
Keywords: EUS; pancreatic cancer; cytology; fine needle aspiration
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Twisted Syringe (Experimental): briefly disconnecting the syringe from the biopsy channel after a specimen is obtained and then reconnecting it
  Interventions: Other: Twisted Syringe
- Conventional Technique (Active Comparator): syringe is exchanged for the needle stylet and negative pressure is applied allowing acquisition of a cytology specimen.
  Interventions: Other: Conventional Technique

INTERVENTIONS:
Other: Twisted Syringe — briefly disconnecting the syringe from the biopsy channel after a specimen is obtained and then reconnecting it
  Arms: Twisted Syringe
Other: Conventional Technique — syringe is exchanged for the needle stylet and negative pressure is applied allowing acquisition of a cytology specimen.
  Arms: Conventional Technique

SUMMARY:
Endoscopic ultrasound and fine needle aspiration are useful tools for the diagnosis and staging of pancreatic cancer. One potential limitation is contamination when needle traverses the gastrointestinal tract under continuous negative pressure. Gastrointestinal tract contamination can lead to misinterpretation of FNA specimens. We propose a technique to eliminate any remaining negative pressure during EUS-FNA and therefore decrease gastrointestinal tract contamination. Our hypothesis is that briefly untwisting the syringe from the biopsy channel after a specimen is obtained eliminates any remaining negative pressure in the FNA needle and therefore reduces GI tract contamination of EUS-FNA specimens, and will lead to improved diagnostic accuracy of this important clinical technique.

DETAILED DESCRIPTION:
Endoscopic ultrasound (EUS) has evolved into a minimally invasive diagnostic and staging method. The addition of fine needle aspiration (FNA) increases the accuracy of EUS in the diagnosis and staging of pancreatic malignancies. An ultrasound probe attached to the end of the endoscope allows real-time direct visualization by means of ultrasound transmission. During the FNA process a needle is advanced through the biopsy channel of the endoscope and into the target lesion. In order to obtain a tissue specimen of a suspicious pancreatic lesion, an FNA needle must traverse either the stomach or duodenum to access the pancreatic mass. Once the needle has entered the target lesion a syringe is exchanged for the needle stylet and negative pressure is applied allowing acquisition of a cytology specimen. Negative pressure is released from the syringe and the stop cock is closed to the syringe. However, due to the relatively long length of the needle there is is significant remaining negative pressure at the needle tip. This leads to aspiration of surrounding material including GI mucosal contamination into the needle while removing it from the target lesion.

Contamination of the FNA specimen from gastric or duodenal epithelium can occur with continued negative pressure at the needle tip upon withdrawal of the needle out of the target lesion. While EUS-FNA has a high specificity (96%), sensitivity (87%), and accuracy (94%), gastrointestinal tract contamination can lead to misinterpretation of FNA specimens. Based on clinical experience, we propose a technique to eliminate any remaining negative pressure during EUS-FNA and therefore decreasing gastrointestinal tract contamination.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Not pregnant
* Can give consent
* Patients with suspicious GI lesions in need of tissue diagnosis by means of EUS/FNA

Exclusion Criteria:

* Pregnant
* Age < 18
* Cannot give consent
* EUS not technically possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of FNA biopsy | 1 week
  The efficacy of fine needle aspiration is assessed using on site cytopathologists who are blinded with respect to the study ARM. The efficacy of diagnostic yield from samples obtained using the needle-off technique is directly compared to the diagnostic yield of samples obtained using conventional technique.

CONTACTS AND LOCATIONS:
Overall Officials: Kulwinder Dua, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Mitsuhashi T, Ghafari S, Chang CY, Gu M. Endoscopic ultrasound-guided fine needle aspiration of the pancreas: cytomorphological evaluation with emphasis on adequacy assessment, diagnostic criteria and contamination from the gastrointestinal tract. Cytopathology. 2006 Feb;17(1):34-41. doi: 10.1111/j.1365-2303.2006.00277.x. PMID 16417563
- [Derived] Aadam AA, Oh YS, Shidham VB, Khan A, Hunt B, Rao N, Zhang Y, Tarima S, Dua KS. Eliminating the Residual Negative Pressure in the Endoscopic Ultrasound Aspirating Needle Enhances Cytology Yield of Pancreas Masses. Dig Dis Sci. 2016 Mar;61(3):890-9. doi: 10.1007/s10620-015-3860-0. Epub 2015 Sep 7. PMID 26346997